CLINICAL TRIAL: NCT02762864
Title: Post-operative Treatment of Diabetic Peripheral Arterial Disease Guided by Platelet Reactivity Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chi-Hsiao Yeh, MD PhD, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG2F0161
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Peripheral Artery Disease
Keywords: aspirin; ticagrelor; clopidogrel
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Platelet Count; Receptors, Purinergic P2Y12; Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRU-guided (Experimental): dual antiplatelet therapy with clopidogrel 75 mg and aspirin 100 mg daily will be continued for 6 months after the procedure for patients with PRU <234 seconds and followed with single antiplatelet therapy with clopidogrel 75 mg daily throughout the follow-up period. For patients in the PRU-target group with PRU ≥234 seconds, rescue medicine (ticagrelor) will be added to keep PRU<234 seconds.
  Interventions: Other: platelet (P2Y12) reaction units; Drug: ticagrelor; Drug: Comparator
- non PRU-guided (Active Comparator): dual antiplatelet therapy with clopidogrel 75 mg and aspirin 100 mg daily will be continued for 6 months after the procedure for patients with PRU <234 seconds and followed with single antiplatelet therapy with clopidogrel 75 mg daily throughout the follow-up period, regardless the levels of PRU.
  Interventions: Other: platelet (P2Y12) reaction units; Drug: Comparator

INTERVENTIONS:
Other: platelet (P2Y12) reaction units — VerifyNow P2Y12 assay point-of-care testing
Drug: ticagrelor — Antiplatelet therapy approved for ACS. Antagonist of P2Y12 and inhibitor of adenosine diphosphate (ADP)-induced platelet aggregation.
  Other Names: Brilinta
  Arms: PRU-guided
Drug: Comparator — dual antiplatelet therapy with clopidogrel 75 mg and aspirin 100 mg daily will be continued for 6 months after the procedure for patient followed with single antiplatelet therapy with clopidogrel 75 mg daily throughout the follow-up period.
  Other Names: Aspirin; Clopidogrel

SUMMARY:
To compare the effect of PRU(platelet (P2Y12) reaction units)-guided treatment on the change in

1. time of initial leg pain and time of termination of exercise test by pain, evaluated on the graded stationary bicycle test,
2. the lower limb perfusion by using MRI blood oxygenation-level dependent (BOLD) and dynamic contrast enhancement sequences and measures the extracellular volume fraction (ECV) as an indicator of fibrosis severity in calf muscles, from one to 52 weeks post-revascularization in patients with peripheral artery disease who have undergone endovascular revascularization -/+ bypass surgery for moderate to severe claudication or ischemic rest pain.

DETAILED DESCRIPTION:
Patients will be randomly assigned to PRU-guided and non-PRU-guided group. In the non-PRU -target group, dual antiplatelet therapy with clopidogrel 75 mg and aspirin 100 mg daily will be continued for 6 months after the procedure for patient followed with single antiplatelet therapy with clopidogrel 75 mg daily throughout the follow-up period. In the PRU-target group, dual antiplatelet therapy will be the same protocol as in the non-PRU-target group for patients with PRU <234 seconds. However, for patients in the PRU-target group with PRU ≥234 seconds, rescue medicine will be added to keep PRU<234 seconds.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study specific procedures.
2. Ambulatory male or female outpatients with diabetes mellitus aged 18-75 years of age or older at the time of the Screening Visit.
3. Diagnosis of PAD confirmed by history and any one of the following observed in the index (intervention) leg at the Screening Visit:

   1. Resting ABI ≤0.90, or
   2. In patients with an ABI > 1.40 (non-compressible vessels) a resting GTI <0.70 can be used for inclusions.
4. endovascular +/- bypass surgery for superficial femoral artery and/or popliteal and/or tibial arteries, that is planned to occur within 6 weeks after the screening visit. Patients receiving concomitant iliac artery endovascular procedures may be enrolled as long as their procedure also includes treating the distal SFA, popliteal or tibial arteries. The patient is randomised after revascularization procedure has been confirmed as technically successful.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Isolated iliac and/or common femoral arteries lesion.
3. Participation in other clinical study with an investigational product within the last 3 months or any new clinical trial during the course of this study.
4. Gangrene or ischemic ulcer of either lower extremity.
5. PAD of a non-atherosclerotic nature.
6. Chronic oral or parenteral anticoagulant therapy (greater than 7 days)
7. Any health status that would interfere with exercise performance or prevent the patient from completion of MRI examinations.
8. Any major lower limb amputation (minor toe amputations allowed if it does not interfere with ambulation).
9. Myocardial infarction or stroke in the previous 3 months.
10. Any concomitant disease process with a life expectancy of less than 1 year or which is sufficiently severe as to compromise the validity of test performance.
11. Not fully understanding of information pertinent to study conduct or compliance to study procedures.
12. Inability of the patient to comply with study procedures and/or followup (e.g., alcohol or drug abuse).
13. A known bleeding diathesis, hemostatic or coagulation disorder, or systemic bleeding, whether resolved or ongoing.
14. MRI examination is prohibited due to renal insufficiency or renal failure requiring dialysis. Any condition that can not receiving MRI examination, such as claustrophobia, previous abdominal aortic stent(strong artifact).
15. History of previous intracranial bleed at any time, gastrointestinal bleed within the past 6 months, or major surgery within 30 days (if the surgical wound is judged to be associated with an increased risk of bleeding).
16. Hypersensitivity to ticagrelor, aspirin or clopidogrel.
17. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Peak exercise time | month 0,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the leg peak exercise time over time (pre-revascularization and 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.
Limb hemodynamics (Ankle Brachial Index or Great Toe Index) | month 0,1,6,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the Limb hemodynamics (Ankle Brachial Index or Great Toe Index) over time (pre-revascularization and at 1, 6, and 12 months post-revascularization) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.
leg pain MRI perfusion measures | month 0,4,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the lower leg muscle GOLD perfusion measure over time (pre-revascularization, 4, and 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.
Quality of life measures | month 0,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the quality of life over time (pre-revascularization and 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.

SECONDARY OUTCOMES:
Major lower leg events (above the ankle amputations, revascularization procedures) | month1, 3, 6,9,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the major lower limb events, including above ankle amputation, new ulceration, and revascularization procedures over time (pre-revascularization and 1, 3, 6, 9, 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.
Major bleeding events | month1, 3, 6,9,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in bleeding events analyzed using the Thrombolysis in Myocardial Infarction Study Group (TIMI), PLATO, Bleeding Academic Research Consortium (BARC) and International Society of Thrombosis and Haemostasis (ISTH) definitions over time (pre-revascularization and 1, 3, 6, 9, 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.
leg pain (claudication) onset time | month 0,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the leg pain (claudication) onset time over time (pre-revascularization and 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.
Major cardiac events (myocardial infarctions, admission due to congestive heart failure and strokes, and death) | month 1, 3, 6,9,12,or Early Termination
  To compare the effects of PRU-guided versus non-PRU-guided treatment on changes in the major cardiac events including fatal and non-fatal myocardial infarctions, admission for congestive heart failure, and strokes, and death over time life over time (pre-revascularization and 1, 3, 6, 9, 12 months post-revascularization, or early termination ) during 12 months of therapy in patients with Peripheral Artery Disease who have undergone endovascular -/+ bypass surgery revascularization for moderate to severe claudication or ischemic rest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hsiao Yeh, MD pHD, Principal Investigator — Chang Gung Memorial Hospital, Keeln\ung